CLINICAL TRIAL: NCT06765226
Title: Abiomed Impella Pump Return Registry - Observational Study
Brief Title: Impella Pump Return Study to Analyze Deposits and Biomaterial in Used Pumps
Status: Recruiting | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-R01
Record Dates: First submitted 2025-01-02; First posted 2025-01-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Impella CP: Patients treated with Impella CP heart pump for more than 4 days due to severe acute heart failure by any cause
- Impella 5.5: Patients treated with Impella 5.5 heart pump for more than or equal to 25 days due to severe acute heart failure by any cause

SUMMARY:
Analysis of cell and protein deposits on the Impella Heart Pump.

DETAILED DESCRIPTION:
The Impella heart pump supports patients in cardiogenic shock for various reasons and has passed safety and biocompatibility evaluations. The planned investigation aims to further analyze cell and protein adhesion on these pumps and the effects of their prolonged use, especially in scenarios like bridge-to-transplant, recognizing preclinical testing limitations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Impella 5.5 therapy and duration of support for ≥ 25 days OR Patients with Impella CP therapy and duration of support for > 4 days

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Impella CP or Impella 5.5 heart pump due to severe acute heart failure by any cause (e.g. cardiogenic shock in acute myocardial infarction, cardiac arrest, myocarditis or in relation to cardiac surgery).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-21 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Investigate deposits and biomaterial after use of pump | through study completion, at least 5 days
  investigate Impella CP after use regarding deposits and biomaterial
Investigate deposits and biomaterial after use of pump | through study completion, at least 25 days
  investigate Impella 5.5 pumps after use regarding deposits and biomaterial

SECONDARY OUTCOMES:
Relation deposits and biomaterial to clinical events | through study completion, at least 5 days
  By correlating patient data, such as medical history and Impella CP related blood parameters, with the findings from our pump analysis, potential connections between medication, diseases, comorbidities, and deposits on the pump can be identified.
Relation deposits and biomaterial to clinical events | through study completion, at least 25 days
  By correlating patient data, such as medical history and Impella 5.5 related blood parameters, with the findings from our pump analysis, potential connections between medication, diseases, comorbidities, and deposits on the pump can be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Lanmüller, MD, Principal Investigator — Deutsches Herzzentrum der Charité
Locations (7):
- Germany (7):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Herzzentrum Dresden, Dresden, Saxony
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Deutsches Herzzentrum der Charité Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Westdeutsches Herz- und Gefäßzentrum Essen, Essen

IPD SHARING:
Plan to Share IPD: Undecided
No publication planned yet